CLINICAL TRIAL: NCT00080028
Title: Phase I Trial of Motexafin Gadolinium and Chemoradiation in Locally Advanced, Squamous Cell Carcinoma of the Head and Neck
Brief Title: Motexafin Gadolinium With Chemotherapy and Radiation Therapy for the Treatment of Advanced Head and Neck Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0210
Record Dates: First submitted 2004-03-22; First posted 2004-03-23 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-05

CONDITIONS: Head and Neck Cancer; Oropharynx Cancer; Larynx Cancer; Hypopharynx Cancer
Keywords: Head and Neck Cancer; SCCHN; Oropharynx Cancer; Hypopharynx Cancer; Larynx Cancer; Soft palate Cancer; Tonsil Cancer; Base of tongue Cancer; Supraglottic Cancer; Glottic Cancer; Pyriform Sinus Cancer; Pharyngeal wall Cancer; Throat cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Hypopharyngeal Neoplasms; Tonsillar Neoplasms | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: Motexafin Gadolinium Injection

SUMMARY:
The purpose of this study is to evaluate the safety of adding the investigational drug Motexafin Gadolinium to the standard treatment of radiation therapy and chemotherapy with drugs called 5-FU and cisplatin in patients with advanced head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Each patient must sign a study-specific informed consent form
* Newly diagnosed, locally advanced, non-metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN) arising from a primary site in the oropharynx, hypopharynx, or larynx confirmed by evaluation of fine needle aspiration or biopsy samples and MRI
* Eligible for curative intent treatment with hyperfractionated radiation and concurrent 5-FU and cisplatin
* Karnofsky Performance Status score of at least 60%
* Primary tumor at least 4 cm in diameter

Exclusion Criteria:

Laboratory Values of:

* Serum creatinine > 1.8 mg/dL; unless 24-hour urine creatinine clearance is ≥ 70 mL/min
* Serum total bilirubin > 1.5 times the upper limit of normal
* ALT (formerly SGPT) > 1.5 times the upper limit of normal
* Alkaline phosphatase > 1.5 times the upper limit of normal
* Absolute neutrophil count (ANC) < 1500/L
* Platelet count < 100,000/L
* 3+ or greater proteinuria on urinalysis

and

* Squamous Cell Carcinoma of the Head and Neck arising from a primary site in the oral cavity or nasopharynx
* Distant metastases
* Prior history of cancer at any site treated with radiotherapy and/or chemotherapy
* History of SCCHN diagnosed within 5 years of current diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - University of Texas, San Antonio Health Science Center, San Antonio, Texas